CLINICAL TRIAL: NCT04813601
Title: Estudio Piloto de Una Serie de Casos Para Evaluar el Efecto Rehabilitador Del Uso de un Exoesqueleto de Marcha en Pacientes Con patología Neuromuscular o parálisis Cerebral
Brief Title: Rehabilitative Effect of the Use of a Gait Exoskeleton in Patients With Neuromuscular Disease or Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MarsiBionics (Industry)
Collaborators: Hospital Universitario La Paz (Other); National Research Council, Spain (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATLAS2030CLI-I
Record Dates: First submitted 2021-03-15; First posted 2021-03-24 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Neuromuscular Diseases; Cerebral Palsy; SMA II
Keywords: Gait Exoskeleton; Robotics; Children; ATLAS 2030; Neuromuscular disease; Cerebral Palsy; Rehabilitation
MeSH Terms: conditions — Neuromuscular Diseases; Cerebral Palsy; Spinal Muscular Atrophies of Childhood

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Robot Asissted Gait Training (Experimental): The rehabilitation sessions will be carried out by a physiotherapist trained in rehabilitation with the ATLAS 2030 exoskeleton and will also have the technical supervision of personnel specialised in the handling of the laboratory and the robotic device.
  Interventions: Device: ATLAS 2030

INTERVENTIONS:
Device: ATLAS 2030 — The participant will attend the laboratory every week, two days a week. The therapy will consist of the use of the exoskeleton for rehabilitative purposes. At the end of each three-month period, each patient's data will be monitored.
  Other Names: Robot Asissted Gait Training

SUMMARY:
The purpose of this multicentric study is to assess the rehabilitative effect derived from the use of the ATLAS exoskeleton in children with neuromuscular diseases or cerebral palsy and with a level of less than 3 or less in the Functional Ambulation Classification (FAC) as a consequence of their disease, as well as the assessment of other physical, functional and quality of life parameters of interest. For this purpose, the exoskeleton will be used as a rehabilitation and walking assistance tool.

Before starting the study programme and if deemed necessary, a preliminary phase consisting of 1 to 3 sessions will be carried out during which the patient will be shown the exoskeleton for the first time and it will be considered whether any improvements to the different parts of the device or the software are necessary to increase the ergonomics and comfort of the patient.

DETAILED DESCRIPTION:
The objectives of the study are:

* Objective 1: To assess the safety and physical and physiological tolerance of the child to the activity performed with the exoskeleton in the rehabilitation sessions.
* Objective 2:
* To assess the safety of a progressive treatment algorithm to achieve the safe progression of patients throughout the therapy
* To assess whether an improvement is achieved in parameters related to the physical rehabilitation of the patient using the exoskeleton, in respiratory capacity, self-perceived quality of life (physical and emotional well-being and self-esteem) as well as to assess the effectiveness of a psychological intervention to provide support in coping with the situation of using the device for the first time in those children who have not used it before.

The time period of the study will be as long as necessary to reach the desired number of participants, in this case 10 children (N=10). The participants will be patients affected by neuromuscular diseases or cerebral palsy and will be selected on the basis of the following inclusion/exclusion criteria:

Inclusion criteria: 1. Children with neuromuscular disease or cerebral palsy who present gait disturbances or no gait disturbance. 2. Children between 3 and 11 years of age.

Exclussion criteria: not fulfil the usage criteria of the device.

ELIGIBILITY:
Inclusion Criteria:

* Children with neuromuscular disease or cerebral palsy who have gait disturbance or no gait.
* Children between 3 and 14 years of age.

Exclusion Criteria:

* Weight> 35 kg
* Femoral length (from the axis of the hip joint in the sagittal plane to the axis of the knee joint in the same plane) <23 cm or >38 cm for size M and from 31 cm to 40 cm for size L
* Stem length (from the axis of the knee joint in the sagittal plane to the axis of the ankle joint in the same plane) <23 or >32 cm for size M and from or >39 cm for size L
* Distance between great trochanters <24 or >35 cm for size M and <25 cm or >35 cm for size L
* Inability to understand simple commands, to cooperate actively in therapy, or inability to express basic needs
* Spasticity measured with the Modified Ashworth Scale greater than or equal to 3 in the lower limbs
* Scoliosis > 25° without the possibility of wearing a brace
* Skin alteration where direct contact between the patient's skin and the exoskeleton is not recommended
* Limitation of passive range of motion at the knee or hip joint > 20 degrees
* Osteoporosis that may induce a bone fracture when low intensity physical activity is performed
* Any other medical condition that may be a risk to the patient's safety and well-being in relation to low intensity physical exercise

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2020-03-09 (Actual); Primary Completion 2021-03-09 (Actual); Study Completion 2023-09-24 (Actual)

PRIMARY OUTCOMES:
Muscular balance | 1 month
  Strength measured in Newtons with a Hand-Held Dinamometer for elbow flexion, neck lateralization, ankle plantarflexion and dorsiflexion, knee flexion and extension.
Expanded Hammersmith Functional Motor Scale | 3 months
  Motor functionality measured for children with Spinal Muscular Atrophy
Gross Motor Function Measure 88 (GMFM-88) | 3 months
  Motor functionality measured for children with Cerebral Palsy.
Respiratory rate | 1 day
  Respiratory rate measured manually in breaths per minute using chronometer
Heart rate | 1 day
  Measured in beats per minute using vital sign monitor
Oxigen Saturation | 1 day
  Measured in %O2 using vital sign monitor
Blood preasure | 1 day
  measured in mmHg with a sphyngomanometer
Respiratory functional parameters | 3 months
  Measured by Spirometer (volumes measured in litres and pressures in mmHg)
Quality of life assessment | 3 months
  Quality of life iof the children measured using the KINDL questionnaire.
Joint range of motion | 1 month
  Range of motion in degrees of hip, knee and ankle movements using a manual goniometer.
Revised Upper Limb Module (RULM) | 3 months
  Upper limb quality of movement using RULM scale for Spinal Muscular Atrophy children
Quality Upper Extremity Skill test (QUEST) | 3 months
  Upper limb quality of movement using QUEST scale for cerebral palsy children
The Functional Independence Measure for Children (WeeFim) | 3 months
  WeeFim scale for CP children.
Egen Klassifikation | 3 months
  Functional ability measured using EK2 scale for SMA
Skin integrity | 1 day
  Skin alterations assessing their localization, size (centimeters), redness and temperature increase.
Fatigue | 1 day
  Patient fatigue measured by Borg fatigue scale for children ages
Pain assessment | 1 day
  Patient pain measured by EVA faces scale for children ages
Peak Flow cough | 1 week
  Measured in litres per minute using a Peak flowmeter

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Espinosa García, Medicine, Principal Investigator — Hospital Universitario La Paz
Locations (1):
- MarsiCare, Arganda, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: starting 6 months after publication
Access Criteria: Researchers who will asked for this data and with previous approval provided by reserach sponsor